CLINICAL TRIAL: NCT07014566
Title: Effectiveness of Digital Physiotherapy in the Short and Long-Term Management of Lower Extremity Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Selva Otsay, Principal Investigator, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lenfödemalt2025
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2019-02

CONDITIONS: Lower Extremity Lymphedema
Keywords: Lower extremity lymphedema; Digital physiotherapy; Combined decongestive therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Combined Decongestive Therapy Group (Experimental): Patients received digital combined decongestive therapy, including self-bandaging, self-manual lymphatic drainage, breathing exercises, and skin care education, with remote supervision over 4 weeks, followed by a maintenance phase with compression stockings.
  Interventions: Other: Digital Combined Decongestive Therapy

INTERVENTIONS:
Other: Digital Combined Decongestive Therapy — The intervention consisted of a digitally delivered combined decongestive therapy (CDT) program for patients with unilateral or bilateral lower extremity lymphedema. Patients attended a single face-to-face session where a physiotherapist provided training on skin care, self-bandaging, self-manual lymphatic drainage, and therapeutic exercises (breathing, gluteal sets, knee sets, and toe movements). Caregivers recorded the demonstrations for home use. Following this session, a 4-week remote physiotherapy program was implemented using telecommunication technologies. Patients continued self-management with guidance via digital platforms. Compression stockings replaced self-bandaging during the 12-week follow-up phase.

SUMMARY:
This study investigated the short- and long-term effects of digital physiotherapy in patients with unilateral and bilateral lower extremity lymphedema. Limb volume and quality of life were assessed at baseline, post-treatment, and 12-week follow-up.

DETAILED DESCRIPTION:
This study evaluated the feasibility and effectiveness of a digital physiotherapy program based on combined decongestive therapy in patients with lower extremity lymphedema. After an initial face-to-face training session on self-bandaging, self-manual lymphatic drainage, breathing exercises, and skin care, patients followed a 4-week digital physiotherapy program with remote supervision. Compression stockings were used during the maintenance phase. Limb volume was measured using circumference method. Quality of life was assessed with the Lymphoedema functioning, disability and health questionnaire questionnaire. Assessments were repeated post-treatment and at 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral lower extremity lymphedema (either primary or secondary)
* Patients aged 18 years or older

Exclusion Criteria:

* Presence of metastatic disease
* History of coronary heart disease, pulmonary disease, or acute infection of any cause
* Presence of peripheral neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Limb Volume | At baseline, at week 4 (end of treatment), and at week 12 (follow-up)
  Limb volume was assessed by measuring the circumference of the affected arm at 4-cm intervals from the ulnar styloid to the axillary region using a standard tape measure. These measurements were used to calculate the total limb volume to evaluate changes after the intervention and at follow-up.

SECONDARY OUTCOMES:
Change in Quality of Life | At baseline, at week 4 (end of treatment), and at week 12 (follow-up)
  Quality of life was assessed using the Turkish version of the Lymphedema Functioning, Disability and Health Questionnaire (Lymph-ICF), which is specific to lymphedema. The scale consists of 29 items across five domains: physical function, mental function, household activities, mobility activities, and social life. Each item was scored on a 0-100 mm visual analog scale (VAS), where higher scores indicate greater impairment and reduced quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu X, Liu Y, Zhu D, Wang F, Ji J, Yan H. Early prevention of complex decongestive therapy and rehabilitation exercise for prevention of lower extremity lymphedema after operation of gynecologic cancer. Asian J Surg. 2021 Jan;44(1):111-115. doi: 10.1016/j.asjsur.2020.03.022. Epub 2020 May 10. PMID 32402630